CLINICAL TRIAL: NCT00325650
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Assess the Efficacy and Safety of Long-term Administration of Rimonabant in the Prevention of Type 2 Diabetes in Patients With Prediabetic Status (i.e., Impaired Fasting Glucose (IFG), Impaired Glucose Tolerance (IGT) or Both)
Brief Title: Rimonabant In Prediabetic Subjects To Delay Onset Of Type 2 Diabetes
Acronym: RAPSODI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC5107
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Prediabetic State
Keywords: Prediabetic state; Impaired fasting glucose; Impaired glucose Tolerance
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily
  Interventions: Drug: Rimonabant
- Placebo (Placebo Comparator): Placebo (for Rimonabant) once daily.
  Interventions: Drug: Placebo (for Rimonabant)

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: Placebo (for Rimonabant) — Tablet, oral administration
  Arms: Placebo

SUMMARY:
Primary objective:

To evaluate the effect of long-term administration of Rimonabant on the time of progression to type 2 diabetes in patients with prediabetes (i.e. Impaired Fasting Glucose (IFG) or Impaired Glucose Tolerance (IGT) or both at baseline).

Secondary objectives:

* To assess the effect on weight loss and weight maintenance; sustained effect following a washout period, effect on other markers of glycemic control (fasting glucose, fasting-insulin and HbA1c), glucose tolerance and insulin responses during oral glucose tolerance tests (OGTTs), and on other risk factors (HDL-Cholesterol, TG),
* To assess the effect on quality of life
* To evaluate long term safety and tolerability.

DETAILED DESCRIPTION:
The total duration per patient will be approximately 38 months including a 30-month double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* No previous history of treatment for type 2 diabetes.
* Diagnosis of :

  * Impaired Glucose Tolerance (IGT) based on one oral glucose tolerance test (OGTT) and defined as a 2 hour post-challenge glucose (after a 75-g Oral Glucose Tolerance Test) > 140 mg/dL (7.8 mmol/L) but < 200 mg/dL (11.1 mmol/L), at the screening visit.
  * And / or impaired fasting glucose (IFG) based on a Fasting Plasma Glucose (FPG) ³ 100 mg/dL (5.6 mmol/L) and < 126 mg/dL (7.0 mmol/L), at the screening visit.

Exclusion Criteria:

* Absence of effective contraceptive method for females of childbearing potential.
* Presence of any clinically significant endocrine disease according to the Investigator.Note: euthyroid patients on replacement therapy will be included if the dosage of thyroxine is stable for at least 3 months prior to screening visit.
* Presence of any severe medical or psychological condition or chronic conditions/infections that in the opinion of the Investigator would compromise the patient's safety or successful participation in the study.
* Presence or history of cancer within the past five years with the exception of adequately treated localized basal cell skin cancer or in situ uterine cervical cancer.
* Related to laboratory findings:

  * positive test for hepatitis B surface antigen and/or hepatitis C antibody;
  * Positive urine pregnancy test in females of childbearing potential ;
  * Thyroid-stimulating hormone (TSH) and free T4 outside central laboratory normal range.
* Related to previous or concomitant medications:

  * Within 3 months prior to screening visit and/or during the screening period:

    * anti-obesity drugs (e.g., sibutramine, orlistat, herbal preparations, etc),
    * systemic long-acting corticosteroids; prolonged use (more than 10 days) of systemic corticosteroids;

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2420 (Actual)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Time of progression to type 2 diabetes | Baseline to 30 months

SECONDARY OUTCOMES:
Change from baseline in body weight | Baseline to 30 months
Change from baseline in waist circumference | Baseline to 30 months
Change from baseline in in glucose homeostasis (HbA1C, fasting plasma glucose and fasting insulin) | Baseline to 30 months
Change from baseline in glucose and insulin at 2 hour post-glucose load | Baseline to 30 months
Change from baseline in HDL-Cholesterol and triglycerides (TG) | Baseline to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States